CLINICAL TRIAL: NCT01254448
Title: Two-Part, Sequential Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TC-5619-238 in Elderly Subjects With and Without Alzheimer's Disease
Brief Title: Multiple Ascending Dose Study of TC-5619 in Healthy Elderly Subjects and Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TC-5619-238-CLP-003
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N-(2-(pyridin-3-ylmethyl)-1-azabicyclo(2.2.2)oct-3-yl)-1-benzofuran-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive a placebo capsule orally once a day for 28 days (Group 1) or 10 days (Group 2).
  Interventions: Drug: Placebo
- TC-5619 (Experimental): Subjects will receive a TC-5619 orally once a day for 28 days (Group 1) or 10 days (Group 2).
  Interventions: Drug: TC-5619

INTERVENTIONS:
Drug: TC-5619 — Group 1: 25 mg TC-5619 administered once daily for 28 days. Group 2: 50-150 mg TC-5619 administered once daily for 10 days.
  Arms: TC-5619
Drug: Placebo — Group 1: matching placebo administered once daily for 28 days. Group 2: matching placebo administered once daily for 10 days.
  Arms: Placebo

SUMMARY:
This is a Phase 1 study to examine the safety, tolerability and pharmacokinetics of TC-5619 in elderly subjects with and without Alzheimer's disease. Group 1 includes elderly subjects with Alzheimer's disease to receive TC-5619 or placebo for 28 days to evaluate safety and tolerability. Group 2 includes healthy elderly subjects in a dose escalation design to receive TC-5619 or placebo for 10 days to evaluate safety, tolerability and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria (Groups 1 & 2):

* Normal body mass index (BMI)
* Non-smoking for a minimum of 3 months
* Subjects must be in reasonably good health, based on medical history, physical examination, vital signs, and ECG.

Group 1 Only:

* Subjects a Mini Mental State Examination score between 12-22, inclusive.
* Diagnosis of probable Alzheimer's Disease according to National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Subjects must have a reliable caregiver.

Exclusion Criteria (Groups 1 & 2):

* Subjects with clinically significant heart disease, pulmonary disease, diabetes, neurologic or psychiatric disease (Group 1 subjects must have Alzheimer's Disease), or any other illness that could interfere with interpretation of study results.
* Subjects with a past or current history of seizures cannot participate.
* Current use of donepezil, rivastigmine or galantamine.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Group 1: screening, Days -14, Day -1, Days 1, 2, 3, 27-33; Group 2: Day -14, Day -1, Days 1 -14
  Number of participants with treatment-emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetic profiles | Group 1: Days 1, 2, 28-32; Group 2: Day 1, 2, 4, 8, 10-14
  Plasma concentrations (pharmacokinetic profiles) of TC-5619-238 over time (Groups 1 & 2) and urine (Group 2) samples after multiple doses
Markers of inflammation in cerebrospinal fluid | Group 1: Days 1, 2, 28-32; Group 2: Day 1, 2, 4, 8, 10-14
  Changes in markers of inflammation in cerebrospinal fluid (Group 1 only)
Markers of inflammation in plasma | Group 1: Days 1, 2, 28-32; Group 2: Day 1, 2, 4, 8, 10-14
  Dose related changes in markers of inflammation in plasma over time (Groups 1 & 2)

CONTACTS AND LOCATIONS:
Overall Officials: George Gerson, MD, Principal Investigator — Comprehensive Phase One
Locations (10):
- United States (10):
  - Collaborative Neuroscience Network, Long Beach, California
  - San Francisco Clinical Research Center, San Francisco, California
  - MD Clinical, Hallandale, Florida
  - Galiz Research, Miami Springs, Florida
  - Comprehensive Phase One, Miramar, Florida
  - Compass Research, LLC, Orlando, Florida
  - Atlanta Center For Clinical Research, Atlanta, Georgia
  - Princeton Medical Institutes, Princeton, New Jersey
  - Community Clinical Research, Austin, Texas
  - Aspen Clinical Research, Orem, Utah